CLINICAL TRIAL: NCT03822156
Title: Clinical Analysis of the Patients With Cavitary Pulmonary Tuberculosis and Endobronchial Tuberculosis in the Private-Public Mix Project for Tuberculosis, Ulsan University Hospital Cohort (PPM-UUH Cohort)
Brief Title: Clinical Analysis of the Patients With Cavitary Pulmonary TB and Endobronchial TB in the PPM-UUH Cohort
Status: Completed | Type: Observational
Sponsor: University of Ulsan (Other)
Collaborators: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Kwang Won Seo, Associate professor, division of pulmonology, dept. of internal medicine, University of Ulsan
Other Study IDs: UUlsan; KCT0003707 (Other: Clinical Research Information Service, Republic of Korea)
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Cavity; Bronchoscopy; Acid Fast Bacilli Infection; Multi-drug Resistant Tuberculosis; Transmission; Insolation
Keywords: Cavitary Pulmonary Tuberculosis; Acid fast bacilli (AFB); Isolation; Endobronchial Tuberculosis; Transmission; Drug susceptible test (DST); Ant-tuberculous agent
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant | interventions — Culture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cavitary Pulmonary Tuberculosis: The patients who are diagnosed with the cavitary pulmonary tuberculosis
  Interventions: Other: Observation of AFB smear/culture
- Endobronchial Tuberculosis: The patients who are diagnosed with the endobronchial tuberculosis
  Interventions: Other: Observation of AFB smear/culture

INTERVENTIONS:
Other: Observation of AFB smear/culture — Observation of the patients from group for their AFB smear/culture results

SUMMARY:
This study is a retrospective cohort study. The purpose of this study is to investigate clinical features of the patients with the cavitary pulmonary tuberculosis (TB) and endobronchial TB from the patients who have been registered in this hospital for treatment and follow-up, as part of the "PPM Project (Private-Public Mix project) for Korean National Tuberculosis Control" introduced in Korea since 2007.

DETAILED DESCRIPTION:
Cavitary pulmonary tuberculosis (TB) is known to remain its Infectivity for a longer period of time than the non-cavitary pulmonary TB, which is usually almost inactivated its infectivity within two weeks after the administration of the anti - TB drugs.

However, there are few studies on this, so it is not known how long the infectivity persists, whether there is a correlation with the number of cavities or the size of the cavities between persistence of infectivity.

Meanwhile, endobronchial TB is known also to be highly infectious, unlike simple pulmonary TB.

It is not known how long infectivity can persist after the administration of anti-TB medication, and whether there is any difference in persistence of infectivity regarding the clinical characteristics of endobronchial TB.

In this study, investigators will analyze the retrospective data analysis of UUH-PPM Cohort, a cohort of PPM project patients in the Ulsan University Hospital (UUH).

The PPM project is a "Private-Public Mix project" for the eradication of tuberculosis from Korea, which the Korean government and private medical institutions have been conducting since 2007.

ELIGIBILITY:
A. Cavitary Pulmonary TB Group

Inclusion Criteria:

1. Aged 18 years and older
2. The patient who has the cavitary pulmonary TB

Exclusion Criteria:

1. Age < 18 years
2. Any Malignant patient
3. Patients with bacterial or viral or fungal pneumonia based on the judgment of the attending physician
4. Patients who had a history of any pulmonary cystic lesion such as infected bulla, bullous emphysema
5. Patients who were diagnosed with pulmonary fungal infection or previous its history or any documented culture of the fungus from a bronchial sample including sputum
6. Patients who were diagnosed with bronchiectasis
7. Patients who were diagnosed with NTM-PD (non-tuberculous mycobacterial pulmonary disease) or any documented culture of NTM from a bronchial sample including sputum
8. Patients who were diagnosed with connective tissue disease such as Wegener's granulomatosis, SLE
9. Patients who were diagnosed with TB destroyed lung
10. Patients who were diagnosed with congenital lung disease such as Congenital Cystic Adenomatoid Malformation (CCAM), pulmonary sequestration
11. Patients who were diagnosed with interstitial lung disease such as Lymphangioleiomyomatosis (LAM), idiopathic pulmonary fibrosis (IPF)
12. Patients who were diagnosed with culture-negative pulmonary TB
13. Patients who did not take anti-TB medication more than twice a week on average
14. Patients who were diagnosed with sarcoidosis
15. Patients who were diagnosed with paragonimiasis
16. Patients who were diagnosed with pulmonary thromboembolism due to excluding pulmonary infarction
17. The patient who did not consent
18. Patients who were diagnosed with MDR/XDR TB through AFB culture

B. Endobronchial TB Group

Inclusion Criteria:

1. Aged 18 years and older
2. The patient who has the endobronchial TB through bronchoscopy

Exclusion Criteria:

1. Age < 18 years
2. Patient who was not consented

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who have been registered in this hospital for treatment and follow-up, as part of the "PPM Project (Private-Public Mix project) for Korean National Tuberculosis Control" introduced in Korea since 2007.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
TLSD | at baseline
  Treatment of anti-TB medication to Last Smear positive Duration
TLCD | at baseline
  Treatment of anti-TB medication to Last Culture positive Duration
ACSD | at baseline
  AFB Culture-Smear positive Dissociation
TCV/RLV | at baseline
  TCV/RLV (Total Cavity[ies] Volume/Total Lung Volume) on enhance CT
TTV/RLV | at baseline
  TTV/RLV (Total TB lesion Volume/Total Lung Volume) on enhance CT

SECONDARY OUTCOMES:
Radiological measure for Tb lesions including cavity size, number | at baseline
  analysis by BioView Duet Workstation (BioView Ltd, Rehovot, Israel) [cavitary pulmonary TB]
Admission Duration | at baseline
  The patients' Hospital admission duration [cavitary pulmonary TB and endobronchial TB]
Isolation Duration | at baseline
  The patients' isolation duration during hospital admission [cavitary pulmonary TB and endobronchial TB]
Hemoptysis /Bronchial artery embolization (BAE) | at baseline
  The patients' history of Hemoptysis /Bronchial artery embolization (BAE) [cavitary pulmonary TB and endobronchial TB]
TB PCR, XPERT | at baseline
  The patients' result of TB PCR, XPERT [cavitary pulmonary TB and endobronchial TB]

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Won Seo, M.D., Ph.D., Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, 877 Bangeojin Sunwhando-ro, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No